CLINICAL TRIAL: NCT01101503
Title: The Metabolic Memorial Effect of Early Intensive Multifactorial Treatment in Diabetes
Brief Title: The Effect of Intensive Multifactorial Therapy on Endothelial Function in Newly Diagnosed Type 2 Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiang Guang-da (Other)
Responsible Party: Sponsor-Investigator, Xiang Guang-da, Director of Endocrinol Dept., Wuhan General Hospital of Guangzhou Military Command
Organization: Wuhan General Hospital of Guangzhou Military Command (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: q9jhrvf3
Record Dates: First submitted 2010-04-06; First posted 2010-04-12 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2010-03

CONDITIONS: Endothelial Dysfunction
Keywords: Newly diagnosed type 2 diabetes; Endothelial dysfunction; Intensive therapy; Metabolic Memorial Effect

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive multifactorial group (Experimental): Intensive multifactorial therapy group receive intensive blood glucose, blood pressure and blood lipids control.
  Interventions: Drug: Intensive multifactorial group
- conventional multifactorial therapy group (Experimental): Conventional multifactorial therapy group receive conventional blood glucose, blood lipids and blood lipids control to the local targets.
  Interventions: Drug: conventional multifactorial therapy group

INTERVENTIONS:
Drug: Intensive multifactorial group — Intensive multifactorial therapy and conventional multifactorial therapy will be taken for 1 year, and then take them together, and give same treatment for 10 years.
  The intensive multifactorial therapy group:
  1. For blood glucose control, target HbA1c >=5.5%and <=6.0%,fasting blood glucose >=5.0 mmol/L and <=6.0 mmol/L, postprandial 2 hour glucose >= 6.0 mmol/L and <= 7.8 mmol/L. The drugs include insulin, oral hypoglycemic agents.
  2. For blood lipids control, target LDL-C < =1.9 mmol/L, triglyceride < =1.5 mmol/L. The drugs include statin and fibrate.
  3. For blood pressure control, target >=120/70 mmHg and <= 130/80 mmHg. The drugs include ACE inhibitor, angiotensin II-receptor antagonist, diuretic, beta-blocker and calcium-channel blocker.
  4. Others, such as aspirin.
  Other Names: Intensive group
  Arms: Intensive multifactorial group
Drug: conventional multifactorial therapy group — Intensive multifactorial therapy and conventional multifactorial therapy will be taken for 1 year, and then take them together, and give same treatment for 10 years.
  The conventional multifactorial therapy group:
  1. For blood glucose control, target HbA1c >6.5%and <=7.0%,fasting blood glucose >6.0 mmol/L and <=7.0 mmol/L, postprandial 2 hour glucose > 7.8 mmol/L and <= 10.0 mmol/L. The drugs include insulin, oral hypoglycemic agents.
  2. For blood lipids control, target LDL-C > 1.9 mmol/L and < =2.5 mmol/L, triglyceride > 1.5 mmol/L and < = 2.5 mmol/L. The drugs include statin and fibrate.
  3. For blood pressure control, target >130/80 mmHg and <= 140/90 mmHg. The drugs include ACE inhibitor, angiotensin II-receptor antagonist, diuretic, beta-blocker and calcium-channel blocker.
  4. Others, such as aspirin.
  Arms: conventional multifactorial therapy group

SUMMARY:
The endothelial dysfunction is the early event in atherosclerosis. The investigator previous study showed that impaired endothelial function exist in newly diagnosed type 2 diabetes. The investigators hypothesize that intensive multifactorial therapy including intensive blood control and intensive hypertension control as well as intensive blood lipids control of 1 year can improve vascular endothelial function. Moreover, the improvement of endothelial function maintains after 5 years or 10 years of intensive multifactorial therapy, called "Metabolic Memorial Effect of improvement of endothelial function".

DETAILED DESCRIPTION:
* We select 1000 patients with newly diagnosed type 2 diabetes. They are divided into two groups, respectively (Intensive multifactorial therapy and conventional multifactorial therapy groups). After those therapy for one year, a 10 years of follow up study will be performed. During this period, we take them together intensive education, and take conventional multifactorial therapy for both of two groups.
* At the beginning (0 year),the end of intensive multifactorial therapy (1 year), 5 years and 10 years, we will measure the endothelium-dependent arterial dilation, endothelium related cytokines such as ET-1, vWF,as well as blood glucose, HbA1c for all of individuals.
* We will compare the endothelial function,endothelium related cytokines such as ET-1, vWF,as well as blood glucose, HbA1c between intensive therapy group and conventional therapy group at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 diabetes,
* Age: 40 >= age <=70 year old,

Exclusion Criteria:

* Type 1 diabetes,
* Mitochondrial diabetes
* Patients with clinical detectable angiopathy,
* Body Mass Index (BMI) > 30 Kg/m2,
* Age < 40, or > 70 years old,
* Malignant neoplasms, renal or liver diseases,
* Smokers
* Known diabetes

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2010-04; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The metabolic memory effect of endothelium-dependent arterial dilation | 10 years
  Before and after intensive multifactorial therapy (one year intensive therapy, HbAic, fasting blood glucose and postprandial 2 hour glucose reach to the targets),endothelial function is measured. The intensive and conventional groups are taken together, and give the same therapy during the follow up of 10 years. The endothelium-dependent arterial dilation is measured during follow up. The aim is that the improvement of endothelial function induced by intensive therapy will exist after 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Guangda, MD.Ph D, Study Director — Wuhan General Hospital
Locations (1):
- Department of Endocrinology, Wuhan, Hubei, China